CLINICAL TRIAL: NCT07192445
Title: Exploring the Usability of Graphic Medicine as an Educational Tool Among Psychology Students
Brief Title: Usability of Graphic Medicine in Psychology Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 96-2022-Hf
Record Dates: First submitted 2025-09-04; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Student Education; Psychology
Keywords: comic book; graphic novel; mental health; university
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graphic Medicine Reading Intervention (Experimental): Participants in this arm read selected excerpts from mental health-themed graphic novels. The materials portray personal experiences of individuals with mental health conditions, their families, and healthcare professionals. The excerpts combine narrative text and visual storytelling to illustrate real-life challenges, coping strategies, and perspectives related to mental health. The reading session is completed individually in a classroom setting.
  Interventions: Other: Reading of Mental Health Graphic Novels

INTERVENTIONS:
Other: Reading of Mental Health Graphic Novels — Participants read carefully selected excerpts from graphic novels focused on mental health. These excerpts integrate written narratives with visual storytelling to illustrate daily life challenges, symptoms, interpersonal relationships, and treatment experiences in mental health contexts. The intervention is conducted individually in a supervised classroom environment. Along with the graphic novel, a guide is provided with questions designed to encourage focused and reflective reading.

SUMMARY:
This study explores the use of graphic medicine-which includes comics, graphic novels, and illustrations-as an innovative educational tool for psychology students learning about mental health. Traditional teaching methods, such as lectures and textbooks, are effective for delivering theoretical knowledge but may not fully capture the complexity of mental health experiences or encourage the empathy needed for future clinical practice. Graphic medicine offers a visual and narrative approach that can make abstract concepts more tangible, encourage active participation in learning, and foster emotional connection.

The primary aim of the study is to evaluate the usability of mental health-themed graphic novels among psychology students. Usability is assessed using the User Experience Questionnaire (UEQ), which measures aspects such as attractiveness, clarity, efficiency, reliability, stimulation, and novelty. Secondary aims include examining changes in students' emotional responses (positive and negative affect), motivation to learn about mental health, enjoyment of reading graphic novels, attitudes toward their use in education, willingness to use them in the future, and perceptions of their validity.

This is a pre-post quasi-experimental study involving psychology students from the University of Málaga. During the intervention, participants read selected excerpts from graphic novels that portray real-life experiences of individuals with mental health conditions, their families, and professionals involved in their care. These narratives aim to bridge the gap between theory and real-life application and evoke empathy.

Before and after the reading activity, students complete self-report questionnaires assessing usability and the secondary variables. Data analysis involves Wilcoxon signed-rank test for paired samples, with Bonferroni correction applied to control for multiple comparisons, and a thematic analysis with Atlas.ti.

ELIGIBILITY:
Inclusion Criteria:

* . Second-year Psychology students studying Psychopathology.

Exclusion Criteria:

* . Students with language barriers.
* . Students with severe reading or comprehension difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Usability | Before and after the intervention (Baseline and one hour later)
  The User Experience Questionnaire (UEQ) is designed to help people reflect on their feelings, impressions, and attitudes associated with the use of a product. It consists of six scales: Efficiency, Perspicuity, and Dependability (pragmatic dimension); Stimulation and Novelty (hedonic dimension); and Attractiveness. It presents 26 items that are evaluated on a scale ranging from -3 to +3, where -3 indicates the most negative response, 0 a neutral response, and +3 the most positive. The results are grouped around six main dimensions, organized into two broad categories: pragmatic quality (which encompasses aspects related to the usability and functionality of the resource) and hedonic quality (linked to the emotional, motivational, and aesthetic dimensions of the experience) (Schrepp, 2015).

SECONDARY OUTCOMES:
Positive and negative affect | Before and after the intervention (Baseline and one hour later)
  The extent to which participants experienced positive (fun, joy, optimism, confidence, gratitude, calm, wonder, happiness, etc.) and negative (stress, fear, irritability, guilt, shame, sadness, hatred, nervousness, shyness, etc.) emotions scored on Likert scales (1-5).
Motivation to learn about mental health | Before and after the intervention (Baseline and one hour later)
  The level of interest, engagement, and willingness of participants to learn about mental health scored on a Likert scale (1-10).
Motivation to read mental health graphic novels | Before and after the intervention (Baseline and one hour later)
  The level of interest and willingness of participants to read mental health graphic novels before and after the intervention scored on a Likert scale (1-10).
Enjoyment of reading mental health graphic novels | Before and after the intervention (Baseline and one hour later)
  The degree to which participants found graphic novels enjoyable, engaging, and satisfactory on a Likert scale (1-10).
Attitudes toward graphic novels | Before the intervention (Baseline and one hour later)
  Participants' perceptions of learning effectiveness, empathy, and content retention when using graphic novels compared to traditional learning methods (e.g., lectures) on a Likert scale (1-10).
Perception of graphic novels in mental health education | After the intervention (One hour later)
  Changes in participants' understanding and conceptualization of graphic novels as educational resources in the context of mental health (yes/no).
Willingness to use mental health graphic novels | Before and after the intervention (Baseline and one hour later)
  The degree to which participants expressed willingness to borrow graphic novels from the Graphic Psychology section of the university library on a Likert scale (1-10).
Content validity of the graphic novels | After the intervention (One hour later)
  The content and format of each graphic novel evaluated on a Likert scale (1 = Does not meet the criterion; 5 = High level of compliance with the criterion) (Escobar-Pérez & Cuervo-Martínez, 2008): a) Comprehensibility: It is presented in a way that the content is easily understood, without confusion or ambiguity; b) Adequacy: It is appropriately tailored to address the selected mental health problem; c) Sufficiency: It includes all essential information to adequately represent the chosen mental health issue; d) Clarity: It is easy to understand, without excessive complexity and using appropriate language; e) Coherence: The narrative and visual elements of the graphic novel remain logical and consistent throughout the story: f) Relevance: The content is directly and significantly linked to the mental health issue addressed; g) Format: The visual structure, typography, and layout of the text in the graphic novel are attractive and functional,.
Reflections | After the intervention (One hour later)
  Open-ended questions: a) Empathy: How did the story make you feel?; b) Application to psychology: How could this content be applied in clinical practice?; c) Visual and narrative representation: What impact have the graphic elements (composition, colors, sizes, facial expressions, etc.) had on your understanding as a reader?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Málaga, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lesinska-Sawicka M. Using graphic medicine in teaching multicultural nursing: a quasi-experimental study. BMC Med Educ. 2023 Apr 17;23(1):255. doi: 10.1186/s12909-023-04223-2. PMID 37069640
- [Background] Williams L, Harstade CW, Anderson N, Deshmukh A, Gayton A, Gott M, Guo P, Nicol J, Tavares T, Waterworth S. Nursing students' reactions to a graphic novel: A multi-national descriptive qualitative study. Nurse Educ Today. 2024 Aug;139:106229. doi: 10.1016/j.nedt.2024.106229. Epub 2024 Apr 25. PMID 38691902
- [Background] Consorti F, Fiorucci S, Martucci G, Lai S. Graphic Novels and Comics in Undergraduate and Graduate Medical Students Education: A Scoping Review. Eur J Investig Health Psychol Educ. 2023 Oct 16;13(10):2262-2275. doi: 10.3390/ejihpe13100160. PMID 37887161
- [Background] Anderson PF, Wescom E, Carlos RC. Difficult Doctors, Difficult Patients: Building Empathy. J Am Coll Radiol. 2016 Dec;13(12 Pt B):1590-1598. doi: 10.1016/j.jacr.2016.09.015. PMID 27888946